CLINICAL TRIAL: NCT01124721
Title: Pilot Testing of Cognitive Training on Academic Task Performance in Children With Attention-deficit/Hyperactivity Disorder
Brief Title: Effects of Cognitive Training on Academic Task Performance in Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: Cog-RAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200816598
Record Dates: First submitted 2010-04-30; First posted 2010-05-17 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: ADHD; Attention
Keywords: Cognitive training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed cognitive training (Experimental): Computerized working memory, attention and cognitive tasks
  Interventions: Behavioral: Cognitive training
- Active placebo (Active Comparator): Cognitive training, however the training does not increase in difficulty, or does so to a minimal degree.
  Interventions: Behavioral: Cognitive training-placebo

INTERVENTIONS:
Behavioral: Cognitive training — Cognitive computerized training for several days per week.
  Other Names: Cogmed
  Arms: Cogmed cognitive training
Behavioral: Cognitive training-placebo — Cognitive training that only minimally increases in difficulty
  Other Names: Cogmed placebo
  Arms: Active placebo

SUMMARY:
Impaired WM is a central deficit in ADHD. A computerized training program, Cogmed, has been shown to increase WM capacity in children with ADHD. It is not known whether the training improves behavior associated with classroom learning, such as remaining on-task and inhibiting off- task behavior. The aim of this study is to utilize ecologically valid measures to investigate training's effect on observable ADHD behavior in conjunction with more standard measures. Subjects will be randomly assigned to a Cogmed versus an active "placebo" condition in which the tasks do not increase in difficulty level in a double-blinded fashion. The effects of the active Cogmed versus placebo computer training will be compared on measures in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 7-14
2. At least average academic and intellectual functioning via parent report.
3. Must have ADHD (by parent report of previous diagnosis or per telephone screening checklist - to be confirmed via interview and ratings)
4. Attentional, hyperactive or impulsive symptoms that interfere with functioning.

Exclusion Criteria:

1. Diagnosis of severe mental illness for example, psychotic, bipolar or major depressive disorder, (by history)
2. Mental retardation (by history)
3. English is not the primary language
4. Family does not have a computer

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Restricted Academic Situations Task | 6 weeks
  Assessment of on-task type behavior while doing a simulated academic task.
Working memory measures | 6 weeks
  Assess memory and working memory functioning on computer and or RA administered tests.
Rating scales | 6 weeks
  Parent and teacher ratings of behavior and attention

SECONDARY OUTCOMES:
Fluency and attention measures | 6 weeks
  Measures of fluency and attentional functioning.
Self-control and executive functioning measures | 6 weeks
  Attention and working memory components can affect delay discounting and self-control measures. This measure will assess for change in behavior and ratings associated with executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Schweitzer, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UCaliforniaDavis MIND Institute, Sacramento, California, United States